CLINICAL TRIAL: NCT05116137
Title: The Impact of Resistance ExerciSe on Muscle Mass in GlioblaSToma Survivors (RESIST)
Brief Title: The Impact of Resistance ExerciSe on Muscle Mass in GlioblaSToma Survivors
Acronym: RESIST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Melanie Keats, Principal Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NSH RESIST Trial
Record Dates: First submitted 2021-10-19; First posted 2021-11-10 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Glioblastoma Multiforme of Brain; Brain Cancer
Keywords: Exercise; Circuit-based resistance training; Intervention; Myopathy; Functional status; Quality of life; Randomized controlled trial
MeSH Terms: conditions — Brain Neoplasms; Motor Activity; Muscular Diseases

STUDY DESIGN:
Intervention Model Description: RCTwith 1:1 allocation to intervention or wait-list control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): 12-week circuit-based resistance exercise
  Interventions: Behavioral: Circuit-based resistance exercise (CRT)
- Wait-list Control (No Intervention): Standard of care wait-list control group

INTERVENTIONS:
Behavioral: Circuit-based resistance exercise (CRT) — CRT is a common training method used to foster aerobic fitness, muscular endurance and strength, as well as neuromuscular adaptations in one workout. CRT is comprised of several sets of different exercises with little rest in between each set.
  Arms: Exercise Intervention

SUMMARY:
Glioblastoma patients are confronted with a debilitating disease associated with a low survival rate and poor quality of life. The goal of this study will be to reach a largely underrepresented population in the exercise literature and explore the role of a tailored circuit-based resistance training program on functional fitness (i.e., ability to carry out tasks of daily living) and associated health outcomes (e.g., quality of life) for GBM patients on active treatment.

DETAILED DESCRIPTION:
PROBLEM: Glioblastoma multiforme (GBM) is the most common brain malignancy accounting for approximately 48% of all brain tumors. GBMs are highly vascular and can cause vasogenic brain edema and mass effect, which can worsen the neurologic symptoms associated with the disease. Corticosteroids (i.e., Dexamethasone; DEX) are the treatment of choice to reduce vasogenic edema and intercranial pressure associated with GBM. However, the use of steroids comes at a cost. High dose steroid therapy and/or long-term use results in muscle myopathy (i.e., muscle weakness) in 10-60% of GBM patients, significantly reducing functional ability as well as quality of life (QOL). Thus, adjuvant therapies are needed to help patients maintain their functional ability and QOL. There is a wealth of evidence to support the use of exercise as an adjuvant therapy to improve functional ability as well as help manage treatment-related symptoms. Resistance training (RT) has been shown to increase muscle mass, strength, and functional ability in aging adults and several cancer populations. While limited, studies in GBM have shown that exercise is safe and feasible for this population and that it can improve functional performance. However, no specific research has been performed to determine whether RT can be successfully used in GBM to prevent or reduce steroid induced muscle myopathy. Therefore, the primary purpose of this study is to establish whether an individualized circuit-based RT program will improve functional fitness for patients on active treatment and receiving steroids.

METHODS: This is a two-armed randomized control trial with repeated measures. Thirty-eight adult (18+ years) patients diagnosed with either primary or secondary GBM who are scheduled to receive standard radiation and concurrent adjuvant Temozolomide chemotherapy post-surgical debulking as well as received any dose of DEX will be recruited through the neuro-oncology clinic and the QEII Cancer Center. Patients will be randomly allocated to a standard of care group (SOC) or SOC+RT group (EX). Those in the SOC group will be advised to maintain an active lifestyle for the 12-week intervention whereas those in the EX group will receive a personalized 12-week circuit-based RT program. This program will consist of 3-4 supervised RT sessions/wk. During each session participants will perform a RT program that is comprised of 3 circuits. Each circuit will include 3 sets of 3 different exercises. Each exercise set will be 1 minute in duration (20 seconds/exercise) with 1 minute of rest between sets. Initial exercise intensity will be light and will increase throughout the program based on the participant's progress. All exercise programs will be designed and supervised by a Clinical Exercise Physiologist (CEP). The primary outcome measure for the study is functional performance which will be assessed using the Short Physical Performance Battery and hand grip strength. Secondary outcome measures will include body composition, aerobic fitness, physical activity levels, general health, QOL, fatigue, and cognitive function. All measures will be assessed pre/post-intervention. Safety and exercise adherence will be assessed throughout the study.

ANALYSIS: Descriptive statistics will be used to describe the population, accrual, program adherence and safety. Outcome data will be analyzed using an intention to treat approach. All participants will be entered into a mixed effects model with participant group assignment (EX, SOC) at randomization and timepoint (pre- and post-test) as fixed factors and participant entered as a random factor. Due to feasibility in recruiting participants in the allotted time, the study will not be fully powered to detect sex-based differences; however, effect sizes associated with the intervention will be calculated and presented separately for each sex.

SIGNIFICANCE: This study will demonstrate the not only is RT safe and feasible for those with GBM, but that it also significantly improves functional status by protecting against myopathy. This will help GBM patients maintain their independence which could lead to marked improvements in QOL.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of either primary or secondary GBM
* received any dose of DEX
* Karnofsky Performance Status (KPS) >70
* English fluency
* physician approval
* willingness to travel to Halifax to participate.

Exclusion Criteria:

* unstable or symptomatic cardiac or pulmonary disease, injury or co-morbid disease that precludes ability to safely exercise
* significant cognitive limitations
* uncontrolled seizures associated with impaired awareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Performance | Baseline to post-intervention (12-week) change
  Short Physical Performance Battery to assess activities of daily living
Grip strength | Baseline to post-intervention (12-week) change
  Measured by handheld dynamometer

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Baseline to post-intervention (12-week) change
  Weight (kg) and height (m) will be used to calculate BMI
Body composition and Muscle Mass | Baseline to post-intervention (12-week) change
  Arm, waist, and calf circumference (cm)
Muscle Mass | Baseline to post-intervention (12-week) change
  Muscle mass and quality - 3T diagnostic magnetic resonance imaging
Aerobic fitness | Baseline to post-intervention (12-week) change
  6 minute walk will be used to calculate aerobic fitness
Physical activity | Baseline to post-intervention (12-week) change
  Godin Leisure Time Physical Activity Questionnaire - Leisure Score Index will be used to calculate self-reported leisure physical activity
Physical, functional, emotional, and social/family quality of Life | Baseline to post-intervention (12-week) change
  Functional Assessment of Cancer Therapy - Brain (FACT-Br) - 50 item scale; total scale score range 0-200; higher scores indicate higher overall QOL
Fatigue | Baseline to post-intervention (12-week) change
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) - 13 item scale; score range 0-52; higher scores indicate less fatigue
Cognitive functioning 1 | Baseline to post-intervention (12-week) change
  Trail making test-b; Time taken to complete each task and number of errors made during each task are recorded and compared with normative data. Time to complete the task is recorded in seconds; the greater the number of seconds to complete the task, the greater the impairment.
Cognitive functioning 2 | Baseline to post-intervention (12-week) change
  Hopkins Verbal Learning Test-Revised for memory; total recall and recognition scores will be calculated
General Health (EuroQol) 5 Dimension - 5 Level | Baseline to post-intervention (12-week) change
  Mobility, self-care, usual activities, pain/discomfort, anxiety/depression (EuroQol-5Dimension-5Level; EQ-5D-5L) - 5 dimensions; higher scores indicate higher problems
General Health (EuroQol) Visual Analog Scale | Baseline to post-intervention (12-week) change
  EuroQol Visual Analog Scale 0-100; lower scores indicate worse health

OTHER OUTCOMES:
Study Feasibility - Participant Accrual | Captured over the 12-week study period
  Participant accrual calculated as % of patients referred divided by number of patients consented to participation
Study Feasibility - Participant Attrition | Captured over the 12-week study period
  Participant attrition calculated as % of patients who complete 12-week study divided by number who withdraw from study
Study Feasibility - Participant Adherence | Captured over the 12-week study period
  Participant program adherence calculated as % of exercise sessions completed divided by total number of available exercise sessions over 12-week intervention
Study safety | Captured over the 12-week study period
  Adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Scott Grandy, PhD, Principal Investigator — Dahousie University and Nova Scotia Health Authority; Mary MacNeil, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keats MR, Grandy SA, Blanchard C, Fowles JR, Neyedli HF, Weeks AC, MacNeil MV. The Impact of Resistance Exercise on Muscle Mass in Glioblastoma in Survivors (RESIST): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 May 4;11(5):e37709. doi: 10.2196/37709. PMID 35507403